CLINICAL TRIAL: NCT04065516
Title: Safety and Efficacy of Antireflux Ablation Therapy (ARAT) at Esophagogastric Junction in Patients With Reflux Disease After Peroral Endoscopic Myotomy (POEM) in Achalasia
Brief Title: ARAT for Reflux Disease After Peroral Endoscopic Myotomy in Patients With Achalasia
Acronym: ARAT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-2019-3601-135
Record Dates: First submitted 2019-07-26; First posted 2019-08-22 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Achalasia; Gastroesophageal Reflux
Keywords: Achalasia; Gastroesophageal Reflux; Argon Plasma Coagulation; Peroral Endoscopic Myotomy
MeSH Terms: conditions — Esophageal Achalasia; Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: A clinical trial will be carried out, including all patients with achalasia, treated by peroral myotomy older than 18 years old, with abnormal acid exposure in the pHmetry test 3 months or more after treatment, who accept the management of ablation with hybrid argon plasma. To whom the ablation will be performed with Hybrid Argon Plasma and its effectiveness will be evaluated by clinical questionnaires, endoscopy and pH measurement at the beginning, 2 months, 6 months and 12 months after the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Argon Plasma Coagulation of the gastroesophageal junction (Experimental): Participants with abnormal acid exposure after peroral endoscopic myotomy for achalasia, will be treated by ablation of the gastroesophageal junction with hybrid argon plasma coagulation
  Interventions: Procedure: ARAT technique

INTERVENTIONS:
Procedure: ARAT technique — After an initial endoscopic evaluation, ARAT technique will be performed with marking, submucosal elevation at esophagogastric junction and then ablation with 100-120w of 270-300 degrees at esophagogastric junction, once the application of the therapy is performed mucosal lavage and immersion technique will be made to corroborate integrity and continuity of the gastrointestinal tract and rule out immediate complications.

SUMMARY:
The peroral endoscopic myotomy for the treatment of achalasia is associated with a higher incidence of gastroesophageal reflux disease compared with Heller's myotomy. Remodeling of the esophagogastric junction with hybrid argon plasma could decrease the passage of gastric or gastroduodenal content into the esophagus.

DETAILED DESCRIPTION:
Achalasia is the inability of the lower esophageal sphincter to relax in the context of dysfunction of esophageal peristalsis. Peroral endoscopic myotomy for the treatment of achalasia has an efficacy above 90%, being comparable with Heller's myotomy. The treatment of achalasia by peroral endoscopic myotomy is associated with a higher incidence of gastroesophageal reflux disease, compared with alternative therapies such as Heller's myotomy or pneumatic dilatation. Hybrid argon plasma at the level of the esophagogastric junction could generate remodeling of this region generating a partial stenosis and thereby decrease the passage of gastric or gastroduodenal content into the esophagus.

A clinical trial will be carried out, including all patients with achalasia, treated by peroral myotomy older than 18 years old, with abnormal acid exposure in the pHmetry test 3 months or more after treatment, who accept the management of ablation with hybrid argon plasma. To whom the ablation will be performed with Hybrid Argon Plasma and its effectiveness will be evaluated by clinical questionnaires, endoscopy and pHmetry measurement at the beginning, 3 months, 6 months and 12 months after the procedure.

Demographic and clinical data will be recorded in a data collection sheet, detailing the reflux questionnaire(GERDQ), Eckardt score, endoscopic findings of esophagitis according to Los Angeles classification and abnormal acid exposure in each evaluation. The data will be condensed into a database for subsequent statistical analysis and publication of results.

ELIGIBILITY:
Inclusion Criteria:

* Achalasia type I, II, III
* Treatment with POEM (Peroral Endoscopic Myotomy)
* Abnormal acid exposure (>6%) in the 24h-pHmetry test more than three months after the procedure
* Signed informed consent

Exclusion Criteria:

* Patients who do not accept the treatment
* Previous antireflux surgery
* Previous Heller's Myotomy
* Hiatal hernia greater than 3 centimeters
* Hill's Classification Grade IV
* Pregnancy
* Patients with any contraindication for an endoscopy
* Patients with esophageal or gastric varices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
A change in erosive esophagitis grade assessed by upper endoscopy after ARAT | measures will be performed at 3,6 and 12 months after ARAT
  Upper endoscopy is going to be used to measure the erosive esophagitis grade using the Los Angeles Esophagitis scale(grade A=mild, Grade B=moderate, Grade C=moderate high and Grade D=severe) after after ARAT
A change in esophageal acid exposure assessed by pHmetry study after ARAT | measures will be performed at 3,6 and 12 months after ARAT
  A 24-hours pHmetry study is going to be used to measure esophageal acid exposure in esophagus after ARAT. DeMeester Score and the percentage of esophagic acid exposure will be used to assess pathologic reflux (>14.73 and > 6%, respectively)
A change in clinical symptoms of reflux disease assessed with a gastroesophageal reflux questionnaire after ARAT | measures will be performed at 3,6 and 12 months after ARAT
  The clinical evaluation of reflux disease is going to be assessed by the use of a clinical gastroesophageal reflux disease questionnaire (GERD-Q) after ARAT. Reflux disease was considered positive when >4 points is observed

CONTACTS AND LOCATIONS:
Overall Officials: Oscar V Hernandez, MD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Centro Medico Nacional Siglo XXI Hospital de Especialidades, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pandolfino JE, Gawron AJ. Achalasia: a systematic review. JAMA. 2015 May 12;313(18):1841-52. doi: 10.1001/jama.2015.2996. PMID 25965233
- [Background] Boeckxstaens GE, Zaninotto G, Richter JE. Achalasia. Lancet. 2014 Jan 4;383(9911):83-93. doi: 10.1016/S0140-6736(13)60651-0. Epub 2013 Jul 17. PMID 23871090
- [Background] Vaezi MF, Pandolfino JE, Vela MF. ACG clinical guideline: diagnosis and management of achalasia. Am J Gastroenterol. 2013 Aug;108(8):1238-49; quiz 1250. doi: 10.1038/ajg.2013.196. Epub 2013 Jul 23. PMID 23877351
- [Background] Akintoye E, Kumar N, Obaitan I, Alayo QA, Thompson CC. Peroral endoscopic myotomy: a meta-analysis. Endoscopy. 2016 Dec;48(12):1059-1068. doi: 10.1055/s-0042-114426. Epub 2016 Sep 12. PMID 27617421
- [Background] Zaninotto G, Bennett C, Boeckxstaens G, Costantini M, Ferguson MK, Pandolfino JE, Patti MG, Ribeiro U Jr, Richter J, Swanstrom L, Tack J, Triadafilopoulos G, Markar SR, Salvador R, Faccio L, Andreollo NA, Cecconello I, Costamagna G, da Rocha JRM, Hungness ES, Fisichella PM, Fuchs KH, Gockel I, Gurski R, Gyawali CP, Herbella FAM, Holloway RH, Hongo M, Jobe BA, Kahrilas PJ, Katzka DA, Dua KS, Liu D, Moonen A, Nasi A, Pasricha PJ, Penagini R, Perretta S, Sallum RAA, Sarnelli G, Savarino E, Schlottmann F, Sifrim D, Soper N, Tatum RP, Vaezi MF, van Herwaarden-Lindeboom M, Vanuytsel T, Vela MF, Watson DI, Zerbib F, Gittens S, Pontillo C, Vermigli S, Inama D, Low DE. The 2018 ISDE achalasia guidelines. Dis Esophagus. 2018 Sep 1;31(9). doi: 10.1093/dote/doy071. PMID 30169645